CLINICAL TRIAL: NCT06527066
Title: Effect of Aromatherapy for Facial Aesthetics in Alleviating Signs of Aging: Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Amanda Karina Santos Vieira, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AVieira
Record Dates: First submitted 2024-07-12; First posted 2024-07-30 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-07

CONDITIONS: Aging Well
Keywords: Aesthetics; Complementary Therapies; Aromatherapy; Nursing
MeSH Terms: interventions — Oils, Volatile

STUDY DESIGN:
Intervention Model Description: G1 will be composed of those whose intervention will only be with the carrier base, the All.me Beauty® Gel Sérum Biocompatível, which serves as a way of diluting the EO and does not interfere with its action and therapeutic process, acting as a placebo. In G2 there will be participants who will receive intervention with geranium EO (Pelargonium graveolens), diluted in All.me Beauty® Gel Sérum Biocompatível, respecting a concentration of 1%, determined based on the work of Sabzghabaee et al. (2011), where tolerability was shown in the application of this 1% EO, on oral mucosa, for the treatment of denture stomatitis; For the present study, the sensitivities of the facial skin and smell were taken into account. The intervention with geranium EO (Pelargonium graveolens) will be made available to G1 after the end of the study protocol, in consideration of the ethical precepts of research involving human beings, according to Resolution nº 466/2012.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind (researcher and statistician), it was not possible to blind the participants, since the geranium EO (Pelargonium graveolens) has a characteristic aroma. The researcher/investigator is also the one who will provide care and evaluate the results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Group (G1) (Placebo Comparator): The Placebo Group (G1) will be composed of those whose intervention will only be with the carrier base, the All.me Beauty® Gel Sérum Biocompatível, which constitutes a way of diluting the EO and does not interfere with its action and therapeutic process, acting as a placebo.
  Interventions: Other: Gel Sérum Biocompatível All.me Beauty®
- Intervention Group (G2) (Experimental): In the Intervention Group (G2) there will be participants who will receive intervention with geranium EO (Pelargonium graveolens), diluted in All.me Beauty® Gel Sérum Biocompatível, respecting a concentration of 1%, determined based on a work where tolerability was shown in the application of this 1% EO, on oral mucosa, for the treatment of denture stomatitis; For the present study, the sensitivities of the facial skin and smell were taken into account.
  Interventions: Combination Product: Geranium (Pelargonium graveolens) essential oil (EO) diluted to 1% in All.me Beauty® Gel Sérum Biocompatível

INTERVENTIONS:
Combination Product: Geranium (Pelargonium graveolens) essential oil (EO) diluted to 1% in All.me Beauty® Gel Sérum Biocompatível — Volunteers must use a total of one gram of the formulation on their face, twice a day, in the morning and at night. The total duration of the protocol will be 12 weeks, with assessment of the participants' skin conditions, in relation to the item "Instrumental Facial Assessment", before treatment and after four, eight and 12 weeks.
  Arms: Intervention Group (G2)
Other: Gel Sérum Biocompatível All.me Beauty® — Volunteers must use a total of one gram of the formulation on their face, twice a day, in the morning and at night. The total duration of the protocol will be 12 weeks, with assessment of the participants' skin conditions, in relation to the item "Instrumental Facial Assessment", before treatment and after four, eight and 12 weeks.
  Arms: Placebo Group (G1)

SUMMARY:
Introduction: aesthetics is one of the specialties for professional nurses and presents a dialogue with Aromatherapy, a practice that uses essential oils (EO) from aromatic plants, being one of the most used integrative therapies for beauty care, youth and well-being. EOs are volatile compounds extracted from the most diverse parts of plants and some, such as geranium (Pelargonium graveolens), have antioxidant action, acting in the regeneration and maintenance of skin tissue, becoming a potential ally in the prevention and/or treatment of wrinkles, as well as general skin aging. Several anti-aging strategies are available, but consumers in aesthetics have increasingly prioritized their health and well-being, desiring non-invasive products and treatments, of natural origin, that guarantee safety and effectiveness. Objective: to evaluate the effect of Aromatherapy in alleviating the signs of aging on the facial skin of women, through a protocol of topical facial application, twice a day, with geranium EO (Pelargonium graveolens) diluted at 1% in Biocompatible Serum Gel All.me Beauty. Method: pilot study with a Randomized Clinical Trial (RCT) design, using the Consolidated Standards of Reporting Trials (CONSORT) as a reference, in its extension to randomized pilot and feasibility trials, double-blind (researcher and statistician). The sample will consist of 38 participants, estimating a loss of 10% throughout the study, who will be randomized between the Placebo Group (G1), whose treatment will be with pure use of the carrier base, and Intervention Group (G2), whose treatment will be with geranium EO diluted to 1% in All.me Beauty® Biocompatible Serum Gel. Participants must perform self-application at home, following a determined protocol and the intervention will respect a standard, in accordance with the guidelines of the manufacturer of the equipment used to measure the participants' progress in terms of wrinkles, hydration and elasticity of the facial skin, these being: Visioscan ® VC 20 Plus, Corneometer® CM 825 and Cutometer® Dual MPA 580.

DETAILED DESCRIPTION:
STUDY

This is a Pilot Study with a Randomized Clinical Trial (RCT) design, using the Consolidated Standards of Reporting Trials (CONSORT) as a reference for reporting the study, in its extension for randomized pilot and feasibility trials, double-blind (researcher and statistician), it was not possible to blind the participants, since the geranium EO (Pelargonium graveolens) has a characteristic aroma.

RECRUITMENT

Participants will be recruited by disseminating the research at the Institute of Integrated and Oriental Therapy, at the School of Nursing of the University of São Paulo and also by snowballing to employees of other units of the university. Interested parties will access a page containing explanatory text with a summary of the study and a link to fill out the Screening Form, prepared via Google Forms, and referring to the exclusion criteria.

For eligible interested parties, an in-person assessment will be scheduled to carry out the topical tolerability test with geranium EO diluted at 1%, in All.me Beauty® Gel Sérum Biocompatível, to be applied to the participant's cubital fossa region, with the aim of to rule out hypersensitivity reactions.

After waiting at least 24 hours for the test to take place, excluding immediate and late reactions, a new face-to-face appointment will be scheduled for those who did not manifest any type of adverse reaction, proceeding with the signing of the Terms of Reference. Free and Informed Consent and full completion of the Clinical Assessment Form, prepared electronically using Research Electronic Data Capture - REDCap Brasil and completed by the researcher using electronic equipment such as a cell phone, tablet or notebook.

The form includes questions pertinent to facial aesthetic treatments, lifestyle habits, clinical history, non-instrumental facial assessment and instrumental facial assessment. In the latter, the condition of the participant's facial skin will be analyzed, in terms of wrinkles, degree of hydration and elasticity, using the instruments Visioscan® VC 20 Plus (wrinkles), Corneometer® CM 825 and Cutometer® Dual MPA 580 (elasticity).

SAMPLE

The sample calculation was carried out based on the result obtained by the R2 parameter of the Cutometer® Dual MPA 580 equipment, which is capable of measuring skin elasticity, achieved in the work of Tumsutti et al., 2021, with a similar design and theme. The sample was sized so that an effect size f = 0.7055230 is detected in an ANOVA model for repeated measures with type I and II errors of 5%. Under these conditions, the minimum sample required is 35 participants in total. Estimating a loss of 10% by the end of the intervention, a total of 38 women will be considered, to be distributed between the Placebo Group (G1) and the Intervention Group (G2).

STUDY LOCATION

All assessments will be carried out by the researcher, in person, in a private office at the Center for Nursing Laboratories in Teaching, Skills, Simulation and Research at School of Nursing of the University of São Paulo.

RANDOMIZATION

An independent statistician will carry out the randomization using a randomized table, generated by a computer program, and identified by a numerical code. The list with the random numbers and names of the participants will be packed in opaque envelopes, numbered and sealed by a professional external to the investigation. The envelopes will be drawn and opened by a third professional external to the research, who will be responsible for distributing each participant into their randomized group.

INTERVENTION

G1 will be composed of those whose intervention will only be with the carrier base, the All.me Beauty® Gel Sérum Biocompatível, which serves as a way of diluting the EO and does not interfere with its action and therapeutic process, acting as a placebo. In G2 there will be participants who will receive intervention with geranium EO (Pelargonium graveolens), diluted in All.me Beauty® Gel Sérum Biocompatível, respecting a concentration of 1%, determined based on a work where tolerability was shown in the application of this 1% EO, on oral mucosa, for the treatment of denture stomatitis; For the present study, the sensitivities of the facial skin and smell were taken into account. The intervention with geranium EO (Pelargonium graveolens) will be made available to G1 after the end of the study protocol, in consideration of the ethical precepts of research involving human beings, according to Resolution nº 466/2012.

Both the geranium EO (Pelargonium graveolens) and its carrier base must present a report describing its components and, in relation to the EO, its degree of purity. The preparation and dilution will be done in a microbiological testing laboratory at School of Nursing of the University of São Paulo and the formulations will be stored in a round plastic bottle with a screw cap, accompanied by a measuring spoon, also made of plastic. The formulation, which must be stored away from light, humidity and heat, will be distributed to participants for self-application at home, following the Application and Storage Protocol.

Volunteers must use a total of one gram of the formulation on their face, twice a day, in the morning and at night. The amount and method of application will be demonstrated at the first meeting and in a video to be prepared by the researcher, which will be sent to the participants. There will be no association with any other technique so that there is no bias in the results obtained.

The type and brand of facial soap for routine home use will be evaluated, as well as the photoprotector, requiring the use of formulations that do not contain anti-aging active ingredients for the face and, in relation to the photoprotector, the additional requirement of not presenting pigmentation, which constitutes as an extra layer of protection.

To minimize or avoid interference in measurements, assessments will respect a pre-established standard: immediately before each assessment, the participant must clean her face with water and neutral liquid soap, provided by the researcher, and then wait 20 minutes at rest. , for acclimatization in a controlled environment with a thermometer and hygrometer to measure environmental temperature and humidity. Assessments will be carried out during the day, at a fixed time and place, under indirect natural lighting and participants will be instructed to appear without makeup.

The total duration of the protocol will be 12 weeks, with assessment of the participants' skin conditions, with regard to the item "Instrumental Facial Assessment", before treatment and after four, eight and 12 weeks, according to thematic and similar drawings. At each in-person assessment and, therefore, once a month during the three months of treatment, the participant will be given a vial unit containing 60 grams of the formulation.

At the end of the intervention, volunteers must respond to a Final Questionnaire, also made with RedCap, where they will be able to explain their impressions regarding the characteristics and performance of the product, such as odor, consistency and effectiveness, in addition to impressions regarding the appearance of the product. own skin.

ASSESSMENT INSTRUMENTS

There are several techniques used in RCTs to evaluate the effectiveness of cosmeceutical treatments, with formulations of plant origin or not, in terms of reducing wrinkles and improving skin hydration and elasticity, and most of them have worked with the following instruments, subject to their updates, which will be made available for this study by the company Tecnotests Produtos e Serviços Ltda.:

Visioscan® VC 20 Plus - Skin topography: assessment of wrinkles in the upper and middle thirds of the face (forehead, eyelid cheek junction and jowls only on the left side of the face). By digitizing the image obtained by a video sensor, it allows the evaluation of the skin surface, obtaining the following clinical parameters: SEr - skin roughness, determined by the presence of dark spots; SEw - number and width of wrinkles, this value being greater or lesser, according to the number of wrinkles; SEsm - skin softness, with a higher value of this variable being an indication of better skin texture and softness; SEsc - skin peeling.

Corneometer® CM 825 - assessment of hydration in the upper and middle thirds of the face (forehead, eyelid cheek junction and jowls only on the left side of the face): its measurement principle is the capacitance of a precision capacitor in a dielectric medium, where changes in the dielectric constant in relation to the variation in hydration of the epidermis, changes the capacitance. The measurement is capable of detecting even the smallest changes in the level of hydration, without being influenced by the deeper layers of the skin, by maintaining its range between 10 and 20 µm from the stratum corneum.

Cutometer® Dual MPA 580 - Skin viscoelasticity: assessment of elasticity in the lower third of the face (forehead, eyelid cheek junction and jowls only on the left side of the face). The measuring principle is based on suction created by negative pressure between the instrument and the skin. The depth of skin penetration is determined by an optical system, composed of a light receptor whose intensity varies according to the depth of suction. The resistance that the skin exerts against suction, due to negative pressure, represents its firmness, and its action of returning to the original position, elasticity, both represented in graphs with curves, also presenting several parameters represented by the letters R, F and Q.

ELIGIBILITY:
Inclusion Criteria:

* cisgender women;
* 45 to 55 years old;
* classification of II and III on the Glogau Scale;
* agree to participate in the research considering the conditions and stages of the study protocol;
* do not present adverse reactions to the topical use of the essential oil and its carrier base.

Exclusion Criteria:

* pregnant women;
* breastfeeding women;
* people diagnosed with neurological, serious dermatological diseases and others serious illnesses;
* people with facial injuries;
* severe allergies or occurrence of serious adverse events due to the use of cosmetics and/or cosmeceuticals in the past;
* participants who present an allergic reaction during the allergenicity test and/or during the study;
* those who underwent aesthetic facial procedures with fillers (except lip fillers) and botulinum toxin up to 6 months before the start of the protocol, PDO threads up to 3 months before, and chemical, mechanical and laser peelings, as well as microneedling, up to 1 month before the beginning of participation;
* use of cosmeceuticals seven to ten days before participating in the study, as well as during it, with only the use of photoprotector being permitted and recommended;
* people who have undergone facial aesthetic surgery, except rhinoplasty.

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Cisgender women
Enrollment: 38 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Facial wrinkles | 12 weeks
  Reduction of facial wrinkles using the Visioscan® VC 20 Plus as an assessment instrument
Facial skin elasticity | 12 weeks
  Improvement of facial skin elasticity using the Cutometer® Dual MPA 580 as a measurement evaluation instrument
Facial skin hydration | 12 weeks
  Increased facial skin hydration using the Corneometer® CM 825

CONTACTS AND LOCATIONS:
Overall Officials: Amanda K S Vieira, Principal researcher, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo Nursing School, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No